CLINICAL TRIAL: NCT05221177
Title: Metabolic Cost of Suspension Exercise Training
Brief Title: Metabolic Cost of Suspension Exercise Training (SET-UTH)
Acronym: SET-UTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SET-UTH
Record Dates: First submitted 2021-12-18; First posted 2022-02-02 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Body Composition; Physical Fitness; Energy Expenditure; Resting Metabolic Rate
Keywords: functional fitness training; bodyweight training; oxygen consumption; resistance training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Participants in this arm will perform six suspension training exercises (acute bout per exercise) at two different conditions (30 and 45 seconds).
  Interventions: Behavioral: TR-30; Behavioral: TR-45
- Control (No Intervention): Participants in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: TR-30 — Suspension training exercises will be performed for 30 seconds and the training volume will be consisted of 1 repetition.
  Arms: Training
Behavioral: TR-45 — Suspension training exercises will be performed for 45 seconds and the training volume will be consisted of 1 repetition.
  Arms: Training

SUMMARY:
In this study, the investigators will be able to estimate the metabolic cost of several foundational suspension training exercises.

DETAILED DESCRIPTION:
Suspension exercise training has become a popular cardiovascular training choice in fitness centers and athletic performance enhancement facilities. Despite widespread use and growing popularity, little is known about the metabolic demands of such a training method. Therefore, the purpose of this study was to quantify the cardiovascular and metabolic cost from various foundational suspension training exercises in order to contribute to a better planning of exercise programs in the real world.

Ten healthy young adults were assigned to execute six suspension training exercises (acute bout) for 30 and 45 seconds. Anthropometric, metabolic, and performance measurements were conducted at baseline. The metabolic cost was estimated from heart rate, blood lactate, resting oxygen uptake, exercise oxygen uptake, and excess post-exercise oxygen consumption measurements using a portable gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years
* Physically active individuals
* Free of chronic diseases
* Free of musculoskeletal injuries
* Nonsmokers

Exclusion Criteria:

* Musculoskeletal injuries
* Chronic diseases
* Use of alcohol, caffeine and any type of ergogenic supplements or medication before (≤6 months) and throughout the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Change in exercise-induced energy expenditure | At pre-exercise, during, and post-exercise session (single bout lasting 30 and 45 seconds)
  Exercise energy expenditure (kcal) will be measured using a portable indirect calorimetry system
Change in excess post-exercise oxygen consumption (EPOC) | At post-exercise session (single bout lasting 30 and 45 seconds)
  EPOC (kcal) will be measured using a portable indirect calorimetry system
Change in blood lactate concentration (BLa) | At pre- and post-exercise session (single bout) at 3 minutes post-exercise
  BLa (mmol/L) concentration will be measured in a microphotometer with commercially available kits.
Change in heart rate | At pre-exercise, during, and post-exercise session (single bout lasting 30 and 45 seconds)
  Heart rate (bpm) will be measured with a wearable heart rate monitor
Change in perceived exertion | At pre-exercise, during, and post-exercise session (single bout lasting 30 and 45 seconds)
  Rating of perceived exertion (RPE) will be measured with the Borg scale (0-10)

SECONDARY OUTCOMES:
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | At baseline
  BMI will be calculated using the Quetelet's equation
Waist circumference (WC) | At baseline
  WC (cm) will be measured using a Gullick II tape
Hip circumference (HC) | At baseline
  HC (cm) will be measured using a Gullick II tape
Waist-to-hip ratio (WHR) | At baseline
  WHR will be calculated by dividing the waist by the hip measurement
Resting metabolic rate (RMR) | At baseline
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Body fat (BF) | At baseline
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
  BF (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass (FM) | At baseline
  FM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat-free mass (FFM) | At baseline
  FFM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Maximal oxygen consumption (VO2max) | At baseline
  VO2max (mL/kg/min) will be assessed by a portable open-circuit spirometry system
Maximal strength (1RM) | At baseline
  1RM (kg) will be measured bilaterally on a horizontal leg press and seated chest press machine..
Muscular endurance | At baseline
  Muscular endurance (repetitions) will be measured on a 1-min curl-up and push-up test.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G. Fatouros, Study Director — University of Thessaly
Locations (1):
- Laboratory of Exercise Physiology, Exercise Biochemistry and Sports Nutrition, School of Physical Education, Sports Sciences and Dietetics, University of Thessaly, Trikala, Greece

REFERENCES:
- [Derived] Chatzikamagianni E, Poulios A, Avloniti A, Rosvoglou A, Liakou C, Papanikolaou K, Stampoulis T, Tsimeas P, Batrakoulis A, Chatzinikolaou A, Draganidis D, Jamurtas AZ, Fatouros IG. Evaluation of the Physiological Responses and Energy Expenditure Induced by Suspension Training Exercises. J Strength Cond Res. 2025 May 16;39(9):933-944. doi: 10.1519/JSC.0000000000005150. PMID 40440526